CLINICAL TRIAL: NCT04449731
Title: Changes in Dietary Behaviours During the COVID-19 Outbreak Confinement in the Adult Population
Brief Title: Changes in Dietary Behaviours During the COVID-19 Outbreak Confinement in the Adult Population (COVIDiet_Int)
Acronym: COVIDiet_Int
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Collaborators: Agricultural University of Athens (Other); University of Zagreb (Other); University of Belgrade (Other); Institute of Technology, Sligo (Other); University of Sarajevo (Other); Lithuanian University of Health Sciences (Other); Jozef Stefan Institute (Other); University of Southern Denmark (Other); Institut Za Javno Zdeavlje (Unknown); University of Skopje (Other); Poznan University of Life Sciences (Other); Bezmialem Vakif University (Other); Unidade Local de Saúde de Coimbra, EPE (Other); Kuwait University (Other); Universidad Nacional de Colombia (Other); Manay Rachna International institute of Research and Studies (Unknown)
Responsible Party: Principal Investigator, Celia Rodríguez Pérez, Associate Professor in Nutrition and Food Science, Universidad de Granada
Other Study IDs: 1526/CEIH/2020
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: Eating behaviours; Mediterranean Diet; COVID-19 confinement; Dietary habits; Physical activity
MeSH Terms: conditions — COVID-19; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult population (> 18 years old): Around 30000 adults (> 18 years old) from 22 different countries.

SUMMARY:
This cross-sectional study will allow to collect eating behaviours data during the COVID-19 confinement, some of them related to the Mediterranean Diet to better understand the eating behaviours of adult population during this novel and exceptional situation.

Hypothesis: The eating habits of the population together with physical activity level will change during the COVID-19 outbreak confinement.

DETAILED DESCRIPTION:
Around thirty thousand adults (18 years old and older) will be recruited from 22 different countries (i.e. including Bosnia and Herzegovina, Colombia, Croatia, Denmark, Egypt, Germany, Greece, India, Ireland, Italy, Kosovo, Kuwait, Lithuania, Montenegro, North Macedonia, Poland, Portugal, Serbia, Slovenia, Spain, Turkey and United Kingdom). A self-administered web-based questionnaire with questions aimed at assessing the dietary behaviours of the adult population during the COVID-19 confinement and before it started, will be distributed using social media and snowball sampling. The questionnaire is based on 44 items including socio-demographic data, MEditerranean Diet Adherence Screener (MEDAS) as a reference of a healthy diet, processed foods intake, changes in their usual food choices and weight gain. All data will be collected online to reach the largest number of participants from all territories.

The main objectives of this study are: 1) to examine whether the COVID-19 outbreak confinement has influenced eating habits among the adult population from the 22 countries previously detailed, and 2) to assess the differences in eating behaviours between the countries involved in the study to have a global overview of the behaviour in the face of confinement that helps in public health decision making related to positive impact on the prevention of chronic diseases and COVID-19-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged from 18 years old and over living in the countries involved in the study.

Exclusion Criteria:

* People under 18 years of age living in countries different from those involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Around 30000 adults from 22 countries including Bosnia and Herzegovina, Colombia, Croatia, Denmark, Egypt, Germany, Greece, India, Ireland, Italy, Kosovo, Kuwait, Lithuania, Montenegro, North Macedonia, Poland, Portugal, Serbia, Slovenia, Spain, Turkey and United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet before and during the COVID-19 confinement | 6 months
  Part of the questionnaire based on the validated PREDIMED MEditerranean Diet Adherence Screener (MEDAS-14). Briefly, one point is scored when the following choices are selected: olive oil for cooking, daily consumption of four or more tablespoons of olive oil, white meat vs. red meat, two or more servings of vegetables, three or more pieces of fruit, less than one serving of red meat, hamburgers, sausages or deli meats, less than one serving of carbonated or sugary drinks, weekly intake of seven or more glasses of wine, three or more servings of legumes, three or more servings of fish/seafood, three or more servings of nuts, less than two servings of non-homemade pastries, white meat such as turkey or chicken preference instead red meat and two or more dishes seasoned with tomato, garlic, onion or leeks and sautéed with olive oil (sofrito).
  The MEDAS-14 score ranges from 0 to 14, whereby higher a scoring reflects greater adherence to the Mediterranean diet.
Eating behaviours | 6 months
  Part of the questionnaire based on changes in frequency of cooking, snacking, alcohol, fast-food intake (higher, lower or similar) and fried foods intake (<1 time a week, 1-3 times a week, 4-6 times a week, 7 or more than 7 times a week, never), type of oil employed for frying (olive oil, sunflower oil or other), number of main daily meals out of home before the confinement (0,1, 2 or 3), difficult finding any type of food (yes/no) or perception of being eating more during the confinement (yes/no).
  In this case, better outcomes are expected if participants increase or maintain the frequency of cooking, use olive oil for frying and decrease or maintain the frequency of snacking, alcohol, fast-food or fried foods intake. Additionally, a good outcome will be considered if participants do not eat more during the confinement and if they do not have problems in finding any type of food.

SECONDARY OUTCOMES:
Level of physical activity during the COVID-19 confinement | 6 months
  The questionnaire includes a question regarding the level of physical activity during the COVID-19 confinement in which the following options are provided: it has increased, it has decreased, it remains as usual, I do not practice physical activity.
  The best outcome will be considered if the participants maintain or increase their physical activity level during the COVID-19 confinement.
Weight gain during the COVID-19 confinement | 6 months
  The questionnaire includes a question about the perception or weight gain during the confinement (increased/decreased/Unknown).
  The best outcome will be considered if the participants do not increase weight during the COVID-19 confinement.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Rodríguez Pérez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodriguez-Perez C, Molina-Montes E, Verardo V, Artacho R, Garcia-Villanova B, Guerra-Hernandez EJ, Ruiz-Lopez MD. Changes in Dietary Behaviours during the COVID-19 Outbreak Confinement in the Spanish COVIDiet Study. Nutrients. 2020 Jun 10;12(6):1730. doi: 10.3390/nu12061730. PMID 32531892
- [Result] Kriaucioniene V, Bagdonaviciene L, Rodriguez-Perez C, Petkeviciene J. Associations between Changes in Health Behaviours and Body Weight during the COVID-19 Quarantine in Lithuania: The Lithuanian COVIDiet Study. Nutrients. 2020 Oct 13;12(10):3119. doi: 10.3390/nu12103119. PMID 33065991
- [Result] Giacalone D, Frost MB, Rodriguez-Perez C. Reported Changes in Dietary Habits During the COVID-19 Lockdown in the Danish Population: The Danish COVIDiet Study. Front Nutr. 2020 Dec 8;7:592112. doi: 10.3389/fnut.2020.592112. eCollection 2020. PMID 33364250
- [Result] Sulejmani E, Hyseni A, Xhabiri G, Rodriguez-Perez C. Relationship in dietary habits variations during COVID-19 lockdown in Kosovo: The COVIDiet study. Appetite. 2021 Sep 1;164:105244. doi: 10.1016/j.appet.2021.105244. Epub 2021 Apr 10. PMID 33848591
- [Result] Pfeifer D, Resetar J, Gajdos Kljusuric J, Panjkota Krbavcic I, Vranesic Bender D, Rodriguez-Perez C, Ruiz-Lopez MD, Satalic Z. Cooking at Home and Adherence to the Mediterranean Diet During the COVID-19 Confinement: The Experience From the Croatian COVIDiet Study. Front Nutr. 2021 Mar 31;8:617721. doi: 10.3389/fnut.2021.617721. eCollection 2021. PMID 33869262
- [Result] Pertuz-Cruz SL, Molina-Montes E, Rodriguez-Perez C, Guerra-Hernandez EJ, Cobos de Rangel OP, Artacho R, Verardo V, Ruiz-Lopez MD, Garcia-Villanova B. Exploring Dietary Behavior Changes Due to the COVID-19 Confinement in Colombia: A National and Regional Survey Study. Front Nutr. 2021 Apr 12;8:644800. doi: 10.3389/fnut.2021.644800. eCollection 2021. PMID 33912582
- [Result] Molina-Montes E, Uzhova I, Verardo V, Artacho R, Garcia-Villanova B, Jesus Guerra-Hernandez E, Kapsokefalou M, Malisova O, Vlassopoulos A, Katidi A, Korousic Seljak B, Modic R, Eftimov T, Hren I, Valencic E, Satalic Z, Panjkota Krbavcic I, Vranesic Bender D, Giacalone D, Bom Frost M, Konic Ristic A, Milesevic J, Nikolic M, Kolay E, Guney M, Kriaucioniene V, Czlapka-Matyasik M, Bykowska-Derda A, Kujundzic E, Taljic I, Brka M, Spiroski I, Cunha Velho S, Patricia Sousa Pinto S, Nascimento Monteiro I, Adriana Pereira J, Dolores Ruiz-Lopez M, Rodriguez-Perez C. Impact of COVID-19 confinement on eating behaviours across 16 European countries: The COVIDiet cross-national study. Food Qual Prefer. 2021 Oct;93:104231. doi: 10.1016/j.foodqual.2021.104231. Epub 2021 Mar 23. PMID 36569642
- [Result] Taljić, I., Brka, M., & Rodríguez-Pérez, C. (2022). Dietary Habits During the COVID-19 Lockdown in Bosnia and Herzegovina's COVIDiet Study. In Central European Congress on Food (pp. 477-485). Springer, Cham.